CLINICAL TRIAL: NCT06917365
Title: Clinical Performance of XPEO-E Liner in SERF Dual-mobility Cups
Acronym: 2024-01-XPEO-E
Status: Not yet recruiting | Type: Observational
Sponsor: Societe dEtude, de Recherche et de Fabrication (Industry)
Responsible Party: Sponsor
Other Study IDs: 2024-A02261-46
Record Dates: First submitted 2025-04-01; First posted 2025-04-08 (Actual); Last update posted 2025-04-23 (Actual); Status verified 2025-04

CONDITIONS: Total Hip Arthroplasty (THA)

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
XPEO-E liner is CE marked under MDD 93/42/CEE by equivalency with CI E liner. No pertaining data on XPEO-E liner is yet available. However, clinical evaluation concludes on a reaching of performance and safety and compliance with essential requirements. This study intends to collect data on XPEO-E in order to allow a transit to MDR 2017/745 (EU).

XPEO-E liner is intended to be used with NOVAE cups and SERF femoral heads and Stems. XPEO-E liner will be used according to their CE marking. These devices are intended for hip replacements with the aim of improving quality of life and reducing pain by replacing a damaged joint.

The follow-up visits are established according to the current practice. Additional procedure will only consist on questionnaires that will be filled by the patient and/or the surgeons.

ELIGIBILITY:
Inclusion Criteria:

* Male or female adults.
* Patient that needs to be implanted with a SERF total hip prosthesis.
* Patient responding to IFU requirement.
* Patient affiliated to French social security.
* Patient who has provided a dated and signed informed consent form.

Exclusion Criteria:

* Patient protected by a French legal measure (under legal protection, guardianship or curatorship).
* Patient unable of expressing consent, according to the investigator.
* Patient deprived of liberty or hospitalized against his consent.
* Pregnant or breastfeeding patient.
* Patient presenting a contraindication to the implantation of medical devices according to the instructions for use.
* Patient with a contraindication to radiographic follow-up.
* Patient not being, a priori, capable of respecting the schedule of follow-up visits, according to the investigator.
* Patient unable to complete a self-questionnaire, according to the investigator.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The target population, with the exception of pregnant or nursing women, consists exclusively of patients who have reached bone maturity (mainly over 65 years of age) with acute pain and/or an ailing joint resulting from a medical condition (mentioned in paragraph "Medical indications") and insufficiently improved by an alternative treatment options, after a period of observation of a few weeks to a few months, and not exhibiting any contraindications (mentioned in paragraph "Contraindications").
  Whatever the medical application, it should be noted that dual mobility cups and liners are particularly appropriate for patients with a high risk of dislocation (serious neurological defects, neuropsychiatric issues, severe neuromuscular deficiencies and dependencies) or with a history of recurring dislocation.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2025-05-01 (Estimated); Primary Completion 2032-03-31 (Estimated); Study Completion 2032-03-31 (Estimated)

PRIMARY OUTCOMES:
Functional improvement | Per operative period to 5 years
  To assess the evolution of patient's functional capacity post-implantation using Harris Hips score (measured from 0 to 100 points, the higher the score the better the outcome)

SECONDARY OUTCOMES:
Survival rate | Per operative period to 5 years
  Calculated using the Kaplan-Meier method
Functional improvement | Per operative period to 5 years
  To assess the evolution of patient's functional capacity post-implantation using HOOS score (40-item questionnaire mesured from 0 to 100, with 100 indicating no symptoms and 0 indicating extreme symptoms )
Functional improvement | Per operative period to 5 years
  To assess the evolution of patient's activity post-implantation using Charnley score
Pain release | Pre operative period to 5 years
  To assess patient's pain (Visual Analogic Scale measured on a scale of 0 to 10 to reflect the intensity of the pain)
Patient's quality of life | Pre operative period to 5 years
  To assess patient's quality of life post-implantation (Forgotten Joint Score mesured from 0 to 100, the higher the score, the less the patient is aware of their affected joint when performing daily activities)
Patient's satisfaction | Post operative period to 5 years
  To assess patients' satisfaction with the operation (4-points question)
Adverse events | Per operative period to 5 years
  To assess the long-term safety of investigational medical devices as well as post-operative safety of the surgery